CLINICAL TRIAL: NCT05482750
Title: Effects of Resistance Training Performed in the Fasted State Compared to the Fed State on Morphological and Neuromuscular Adaptations in Young Adults
Brief Title: Resistance Training in the Fasted State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Eduardo Lusa Cadore, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: URioGrandeESEFID
Record Dates: First submitted 2022-07-25; First posted 2022-08-01 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Fasting; Exercise; Resistance Training
MeSH Terms: conditions — Fasting; Motor Activity | interventions — Resistance Training; Angptl4 protein, mouse

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training in the fasted state (Experimental): Subjects will maintain the standard diet and will perform resistance exercise sessions after overnight fasting (10 to 12 hours). Over the 12 weeks of intervention, participants will perform two sessions a week of resistance exercises.
  Interventions: Other: Resistance training in the fasted state
- Resistance training in the fed state (Active Comparator): Subjects will maintain the standard diet and will perform resistance exercise sessions in the fed state, between 1 and 2 hours after consuming a carbohydrate-containing meal. Over the 12 weeks of intervention, participants will perform two sessions a week of resistance exercises.
  Interventions: Other: Resistance training in the fed state

INTERVENTIONS:
Other: Resistance training in the fasted state — On the first day of evaluations, the subjects will perform the basal metabolic rate (BMR) analysis, as well as familiarization with the neuromuscular tests. After the preliminary tests, the volunteers will perform the pre-intervention procedures. Assessments of body composition, muscle thickness and quality, maximum dynamic strength and maximum power will be performed. In addition, instruments related to dietary control and physical activity level will be applied. Subsequently, in a randomized manner, participants will be allocated to one of two different interventions. During the intervention (8 weeks), the adherence to the standard diet will be verified, as well as body composition, muscle thickness and quality, maximum dynamic strength and maximum power will be reassessed. After the 12 weeks of intervention, the volunteers will perform the evaluations referring to the post-intervention moment, following the same steps of the pre-intervention collections.
  Other Names: Fasting; Strength training
  Arms: Resistance training in the fasted state
Other: Resistance training in the fed state — On the first day of evaluations, the subjects will perform the basal metabolic rate (BMR) analysis, as well as familiarization with the neuromuscular tests. After the preliminary tests, the volunteers will perform the pre-intervention procedures. Assessments of body composition, muscle thickness and quality, maximum dynamic strength and maximum power will be performed. In addition, instruments related to dietary control and physical activity level will be applied. Subsequently, in a randomized manner, participants will be allocated to one of two different interventions. During the intervention (8 weeks), the adherence to the standard diet will be verified, as well as body composition, muscle thickness and quality, maximum dynamic strength and maximum power will be reassessed. After the 12 weeks of intervention, the volunteers will perform the evaluations referring to the post-intervention moment, following the same steps of the pre-intervention collections.
  Other Names: Feeding; Strength training
  Arms: Resistance training in the fed state

SUMMARY:
It is well evidenced in the literature that fasting aerobic exercise generates a series of metabolic differences when compared to exercise performed in the fed state, including the use of fats predominantly as an energy source. Consequently, increases in adaptations to aerobic training, related to health and physical performance, are observed when sessions are performed in the fasted state. In relation to resistance training, the evidence is limited. There is a lack of data in the literature regarding the effects of fasting on resistance exercises and whether this practice may reflect in losses or improvements in morphological and neuromuscular adaptations related to resistance training. Thus, the aim of the present project is to compare the effects of resistance training performed in the fasted state compared to the fed state during 12 weeks on body composition and physical performance in young adults. Thirty-four eutrophic or overweight individuals, not engaged in regular resistance exercises, aged between 20 and 40 years, will be recruited. They will be put on a standard customized diet and will perform 2 weekly sessions of resistance exercise after overnight fasting (10 to 12 hours) or in the fed state, for 12 weeks. Before, in the middle and after this period, evaluations of body composition, muscle thickness and quality, maximum dynamic strength and maximum power will be analyzed. Comparisons will be performed using Generalized Estimating Equations (GEE), adopting the factors group (2 stratifications) and time (3 stratifications). All results will be expressed as mean and standard deviation and the accepted significance level will be 5%.

ELIGIBILITY:
Inclusion Criteria:

* Men and women;
* Aged between 19 and 40 years;
* Body mass index (BMI) between 18 and 29.9 kg/m²;
* Not engaged in regular strength physical exercise (>1 weekly session) for the last 3 months.

Exclusion Criteria:

* Smokers;
* Use of medications and/or supplements that may influence the outcomes evaluated;
* Individuals who have a chronic disease that may prevent physical exercise.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Body mass | 1 minute
  Body mass will be measured using a scale (Urano, Canoas, Brazil).
Lean body mass | 15 minutes
  Lean body mass will be determined using the dual energy X-ray absorption (DEXA) method, using a densitometry machine (Hologic GE, Bedford, USA).
Fat body mass | 15 minutes
  Fat body mass will be determined using the dual energy X-ray absorption (DEXA) method, using a densitometry machine (Hologic GE, Bedford, USA).
Muscle thickness | 30 minutes
  Muscle thickness will be evaluated through ultrasound (Nemio XG, Toshiba, Japan).
Muscle quality | 30 minutes
  Muscle quality will be evaluated through echo intensity of the quadriceps through ultrasound (Nemio XG, Toshiba, Japan).
Maximum dynamic strength | 30 minutes
  Maximum dynamic strength will be assessed using the 1 repetition maximum (1RM) test for bench press and knee extension exercises.
Maximum power | 30 minutes
  The maximum power and the medium power will be evaluated in the bench press and knee extension exercises considering a load of 30 and 70% of 1RM.

CONTACTS AND LOCATIONS:
Locations (1):
- Escola de Educação Física, Fisioterapia e Dança - UFRGS, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided